CLINICAL TRIAL: NCT03732339
Title: Predictive Value of Circulating Tumor Cells in Neoadjuvant Chemotherapy Among Locally Advanced Breast Cancer Patients: a Single-center, Prospective, Exploratory Clinical Trial
Brief Title: CTC in Predicting Neoadjuvant Chemotherapy Among LABC Patients: a Single-center, Prospective, Exploratory Clinical Trial
Acronym: CTCNeoBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Beijing Viroad Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinsong Lu, Chief of Breast Surgery Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-2018-038
Record Dates: First submitted 2018-10-08; First posted 2018-11-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Locally Advanced Breast Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GILUPI CellCollector® (Experimental)
  Interventions: Device: GILUPI CellCollector®

INTERVENTIONS:
Device: GILUPI CellCollector® — Use of GILUPI CellCollector® to detect CTC

SUMMARY:
The GILUPI CellCollector® is the first in vivo CTC isolation product worldwide, which is CE approved. The purpose of this clinical trial is to evaluate the predictive value of CTC in neoadjuvant chemotherapy among locally advanced breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed primary invasive breast adenocarcinoma, anatomic stage T2-4N0-3M0 or T1N1-3M0 before neoadjuvant chemotherapy
* ECOG 0-1
* Adequate organ function
* Consent to undergo CTC analysis in vivo

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Metastatic or recurrent patients
* Uncontrollable infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Predictive value of CTC in ypT0 ypN0 | Change from pre-chemotherapy to 22-28(±7) days after first dose of neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Predictive value of CTC in ypT0, ypT0/is ypN0, near pCR | before and 22-28(±7) days after first dose of neoadjuvant chemotherapy
hypersensitivity | up to 1 year
  Number of participants with hypersensitivity as assessed by CTCAE v4.0
Detection rate of GILUPI CellCollector® | before and 22-28(±7) days after first dose of neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Lu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided